CLINICAL TRIAL: NCT04213248
Title: Effect of Umbilical Mesenchymal Stem Cells Derived Exosomes on Dry Eye in Patients With Chronic Graft Versus Host Diseases
Brief Title: Effect of UMSCs Derived Exosomes on Dry Eye in Patients With cGVHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019KYPJ048
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye
Keywords: Dry eye; UMSC; Exosome; cGVHD
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UMSC-exo treatment (Experimental): Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by UMSC-exo intervention for 2 weeks.
  Interventions: Drug: Umbilical Mesenchymal Stem Cells derived Exosomes

INTERVENTIONS:
Drug: Umbilical Mesenchymal Stem Cells derived Exosomes — Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by UMSC-exo 10ug/drop, four times a day for 14 days. The follow-up visit will be 12 weeks.
  Other Names: UMSC-exo

SUMMARY:
The purpose of this study is to determine whether Umbilical Mesenchymal Stem Cells (UMSCs) derived Exosomes could alleviate dry eye symptoms in patients with chronic Graft Versus Host Diseases (cGVHD).

DETAILED DESCRIPTION:
Among patients with cGVHD, 60% - 90% are affected by dry eye symptoms, presenting as progressive development of dryness, foreign body sensation, photophobia, pain and even blindness, which seriously affect their life quality. At present, the standard first-line treatment of cGVHD is still hormone or combined with immunosuppressant of cyclosporine. The dry eyes related to cGVHD are treated with artificial tears, lacrimal punctum embolization, local immunosuppressant or even blepharoplasty to reduce dry eye symptoms. Although a variety of new immunosuppressants and monoclonal antibodies have been used in clinic, the overall efficacy is still unsatisfactory with apparent side effects, and the period of treatment is long with high-costs. Therefore, it is an urgent task for clinicians to explore new methods of cGVHD related dry eye therapy and improve the survival rate and quality of life of patients.

Exosomes are a kind of membrane vesicles secreted by parental cells, which can mediate the transfer of RNA, protein, DNA and other functional molecules between cells and regulate the function of target cells. The therapeutic potential of UMSC exosomes has been widely studied in diseases of liver, kidney, skin and so on. Previously, we found that UMSC exosomes can significantly alleviate the symptoms of dry eye in the dry eye animal model. At present, we plan to clarify its efficacy in clinical research.

The main objective of this study is to assess the alleviation of dry eye symptoms in patients with cGVHD after UMSC-exo treatment by measuring Ocular Surface Index Score (OSDI), and the second objective include the measurement of tear secretion amount, tear break time, the areas stained by fluorescent, ocular redness, tear meniscus and best corrected visual acuity.

Approximately 27 study subjects will be recruited. The treatment group will receive artificial tears for 2 weeks to normalize the baseline, followed by intervention of UMSC-exo 10ug/drop, four times a day for 14 days. The follow-up visit will be 12-week, progression of dry eye will be measured.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed cGVHD with apparent dry eye symptoms by intern specialists and ophthalmologists, and previous application of artificial tears could not relieve the dry eye symptoms.

And meet the following standards:

1. have the following symptoms in at least one eye: dryness, burning sensation, foreign body sensation, discomfort in the ocular surface or visual fatigue;
2. tear secretion test (Schirmer's Test) of either eye ≤ 10 mm / 5 min;
3. the corneal fluorescein staining score (CFS) was more than 4;
4. Tear break time (TBUT) is less than 10 seconds.

Exclusion Criteria:

1. Those who are allergic to any component of the drug in this study;
2. Pregnant or nursing women;
3. Patients with active fungal, bacterial or viral keratitis or conjunctivitis;
4. have serious heart, lung, liver or kidney diseases;
5. Other incurable ocular diseases before the study; such as glaucoma, uveitis, retinitis pigmentosa.
6. Wearing contact lenses and unwilling to take off in the study;
7. Performed ocular surgery (including cataract surgery) in recent three months;
8. Enrolled in other interventional clinical studies at the same time;
9. Application of eye drops that might affect the clinical study in the past 24 hours;
10. Unable to complete the study according to the investigators' requirements;
11. Serious systemic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2023-05-18 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Ocular Surface Disease Index (OSDI) Score | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  The OSDI is a 12-question validated questionnaire used to measure dry eye symptoms. The OSDI scoring scale ranges from 0 to 100. The lower the score, the more symptomatic relief from dry eye symptoms a patient experiences. Baseline-adjusted scores were tabulated; a decrease over 10 scores from baseline indicates an improvement.

SECONDARY OUTCOMES:
Changes in tear secretion amount by Schirmer's Test | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  The investigator placed a paper strip on the eye under the lower lid for a specified time period. The length of the strip wetted by the tears was measured in millimeters. Baseline-adjusted values were tabulated; a positive number change from baseline indicates an improvement in each eye individually.
Changes in Tear break time | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  time required for dry spots to appear on the surface of the eye after blinking was measured in seconds. Baseline-adjusted scores were tabulated; a positive number change from baseline indicates improvement in each eye individually
Changes in Ocular Surface Staining | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Damage to the ocular surface was assessed using non-toxic ophthalmic dye during slit-lamp review. Corneal and conjunctival staining were graded as per the National Eye Institute (NEI) pictorial scale. The lower the score, the less signs of dry eye disease a patient exhibits. Baseline-adjusted scores were tabulated; a negative number change from baseline indicates an improvement in each eye individually
  Damage to the ocular surface was assessed using non-toxic ophthalmic dye during slit-lamp review. Corneal and conjunctival staining were graded as per the National Eye Institute (NEI) pictorial scale. The lower the score, the less signs of dry eye disease a patient exhibits. Baseline-adjusted scores were tabulated; a negative number change from baseline indicates an improvement in each eye individually
Changes in best corrected visual acuity (BCVA). | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  to understand the effect of exosomes on visual acuity
Changes in conjunctiva redness score | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Description: to explore the effect of exosomes on conjunctiva. Nasal and temporal bulbar conjunctival hyperemia were graded separately in each eye by the investigator under slit-lamp magnification by assigning a score of 0 to 4 for each quadrant based on comparison to the Allergan Dry Eye Redness Scale with photographic reference where: 0=Normal, vessels of bulbar conjunctiva are easily observed; 1=Trace redness; 2=Mild redness; 3=Moderate redness; 4=Severe redness, and each score is associated with a reference photo.
Changes in tear meniscus height | 3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
  Description: to reflect the effect of exosomes on tear production. the distance between the line of reflection along the top of the tear prism to the edge of the eyelid was measured in millimeters. Baseline-adjusted scores were tabulated; a positive number change from baseline indicates improvement. Each eye was assessed individually. Both eyes contributed to the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Xialin Liu, Prof., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Randall Harrell C, Djonov V, Volarevic A, Arsenijevic A, Volarevic V. Mesenchymal Stem Cell-Sourced Exosomes as Potentially Novel Remedies for Severe Dry Eye Disease. J Ophthalmol. 2025 Jan 10;2025:5552374. doi: 10.1155/joph/5552374. eCollection 2025. PMID 39839752